CLINICAL TRIAL: NCT02441712
Title: Supervised Rehabilitation With Patterned Electrical Neuromuscular Stimulation for Patients With Patellofemoral Pain
Brief Title: Rehabilitation With Patterned Electrical Neuromuscular Stimulation for Patients With Patellofemoral Pain
Acronym: PENS for PFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Accelerated Care Plus (Industry); Mid-Atlantic Athletic Trainers' Association (Unknown)
Responsible Party: Principal Investigator, Susan Saliba, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17909
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-10

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motor PENS (Experimental): Motor PENS will be a strong tri-phasic stimulation pattern to the hip, quadriceps, hamstring, and adductors for strength training (50Hz impulses for 200ms every 1500 ms). The stimulus will be administered for 15-minutes followed by the impairment rehabilitation program.
  Interventions: Device: PENS
- Subsensory PENS (Sham Comparator): Subsensory PENS will be a sub sensory stimulus also administered by a tri-phasic stimulation pattern to the hip, quadriceps, hamstring, and adductors (50Hz impulses for 200ms every 1500ms). The stimulus will be administered for 15-minutes followed by the impairment rehabilitation program
  Interventions: Device: PENS

INTERVENTIONS:
Device: PENS

SUMMARY:
This is a Randomized Controlled Trial (RCT) regarding the conservative treatment of patellofemoral pain (PFP) with an impairment based rehabilitation program. Those with PFP can have a variety of impairments, such as knee and hip muscle weakness, poor movement patterns, weak core activation and muscle tightness. Several recent RCT trials have looked at treating single impairments, but to date no RCT have address individualized patient impairments during a rehabilitation program. Abnormal muscle firing patterns have also been identified during functional tasks; such as jogging, stair climbing, and performing a single leg squat. Conflicting studies have produced changes to the quadriceps and hip muscle firing patterns with those with PFP. The abnormal activation patterns has been suggested to be why strengthening programs alone do not improve movement patterns during functional tasks for those with PFP. Patterned electrical neuromuscular stimulation (PENS) is a novel form of electrical stimulation that replicates proper firing patterns based off healthy electromyography patterns. The purpose of the study is to investigate the benefits of PENS with a impairment based rehabilitation program for the treatment of PFP. The rationale for this investigation is to assess the benefits of PENS with therapeutic exercise at improving altered firing patterns of the lower extremity muscles during functional tasks.

ELIGIBILITY:
Inclusion Criteria:

* Insidious onset of symptoms
* Presence of peri- or retro patellar knee pain during at least two of the following functional activities:

Stair ascent or descent, Running, Kneeling, Squatting, Prolonged sitting, Jumping

* Pain for more than 3 months
* Pain >3/10 on VAS
* 85 or less on the Anterior Knee Pain Scale

Exclusion Criteria:

* Previous knee surgery
* Internal Derangement
* Ligamentous instability
* Other sources of anterior knee pain(patella tendonitis, osgood schlatter, knee plica, etc)
* Neurological Involvement
* Any biomedical device
* Muscular abnormalities
* Currently pregnant
* Hypersensitivity to electrical stimulation
* Active infection over the site of the electrode placement

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Assessed by Visual Analog Scale (VAS) | Pain recorded by the VAS will be collected for 4 weeks
  Current and Worse VAS

SECONDARY OUTCOMES:
Changes in Quadriceps Muscle Strength | Up to 4 weeks
  Muscle strength of the quadriceps will be measured by individuals performing a maximum contraction against a small device that will measure force output
Changes in Hamstring Muscle Strength | Up to 4 weeks
  Muscle strength of the hamstring will be measured by individuals performing a maximum contraction against a small device that will measure force output
Changes in Gluteus Medius Muscle Strength | Up to 4 weeks
  Muscle strength of the gluteus medius will be measured by individuals performing a maximum contraction against a small device that will measure force output
Changes in Hip Adductor Muscle Strength | Up to 4 weeks
  Muscle strength of the hip adductors will be measured by individuals performing a maximum contraction against a small device that will measure force output
Changes in Lower Extremity Electromyography during a step down task | Up to 4 weeks
  EMG activity of six lower extremity muscles during a step down task
Changes in Lower Extremity Electromyography during a single leg squat | Up to 4 weeks
  EMG activity of six lower extremity muscles during a single leg squat
Changes in Lower Extremity Electromyography during a lunge | Up to 4 weeks
  EMG activity of six lower extremity muscles during a lunge
Changes in Lower Extremity Electromyography during walking | Up to 4 weeks
  EMG activity of six lower extremity muscles during walking
Changes in Lower Extremity Electromyography during jogging | Up to 4 weeks
  EMG activity of six lower extremity muscles during jogging
Changes in Patient reported outcomes | Up to 4 weeks
  4 patient reported outcomes on pain and function before and after the intervention. These patient reported outcomes are the Anterior Knee Pain Scale, the Activities of Daily Living Scale, the Godin Leisure Scale, and the Fear Avoidance Belief Questionnaire.
Changes in lower extremity kinematics | Up to 4 weeks
  Trunk, hip, knee and ankle movement during the single leg squat, stair ambulation, lunges, walking and jogging
Changes in core strength | Up to 4 weeks
  Trunk endurance will be assessed by front and side plank tasks.
Changes in core activation | Up to 4 weeks
  Core activation will be assessed by real time ultrasound to examine the size of the core muscles

CONTACTS AND LOCATIONS:
Overall Officials: Susan Saliba, PhD, ATC, PT, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Macrum E, Bell DR, Boling M, Lewek M, Padua D. Effect of limiting ankle-dorsiflexion range of motion on lower extremity kinematics and muscle-activation patterns during a squat. J Sport Rehabil. 2012 May;21(2):144-50. doi: 10.1123/jsr.21.2.144. Epub 2011 Nov 15. PMID 22100617
- [Background] Bolgla LA, Boling MC. An update for the conservative management of patellofemoral pain syndrome: a systematic review of the literature from 2000 to 2010. Int J Sports Phys Ther. 2011 Jun;6(2):112-25. PMID 21713229
- [Background] Boling MC, Padua DA, Alexander Creighton R. Concentric and eccentric torque of the hip musculature in individuals with and without patellofemoral pain. J Athl Train. 2009 Jan-Feb;44(1):7-13. doi: 10.4085/1062-6050-44.1.7. PMID 19180213
- [Background] Boling MC, Bolgla LA, Mattacola CG, Uhl TL, Hosey RG. Outcomes of a weight-bearing rehabilitation program for patients diagnosed with patellofemoral pain syndrome. Arch Phys Med Rehabil. 2006 Nov;87(11):1428-35. doi: 10.1016/j.apmr.2006.07.264. PMID 17084115
- [Background] Ferber R, Bolgla L, Earl-Boehm JE, Emery C, Hamstra-Wright K. Strengthening of the hip and core versus knee muscles for the treatment of patellofemoral pain: a multicenter randomized controlled trial. J Athl Train. 2015 Apr;50(4):366-77. doi: 10.4085/1062-6050-49.3.70. Epub 2014 Nov 3. PMID 25365133
- [Background] Ferber R, Kendall KD, Farr L. Changes in knee biomechanics after a hip-abductor strengthening protocol for runners with patellofemoral pain syndrome. J Athl Train. 2011 Mar-Apr;46(2):142-9. doi: 10.4085/1062-6050-46.2.142. PMID 21391799
- [Background] Earl JE, Hoch AZ. A proximal strengthening program improves pain, function, and biomechanics in women with patellofemoral pain syndrome. Am J Sports Med. 2011 Jan;39(1):154-63. doi: 10.1177/0363546510379967. Epub 2010 Oct 7. PMID 20929936
- [Background] Earl JE, Schmitz RJ, Arnold BL. Activation of the VMO and VL during dynamic mini-squat exercises with and without isometric hip adduction. J Electromyogr Kinesiol. 2001 Dec;11(6):381-6. doi: 10.1016/s1050-6411(01)00024-4. PMID 11738950
- [Background] Witvrouw E, Callaghan MJ, Stefanik JJ, Noehren B, Bazett-Jones DM, Willson JD, Earl-Boehm JE, Davis IS, Powers CM, McConnell J, Crossley KM. Patellofemoral pain: consensus statement from the 3rd International Patellofemoral Pain Research Retreat held in Vancouver, September 2013. Br J Sports Med. 2014 Mar;48(6):411-4. doi: 10.1136/bjsports-2014-093450. No abstract available. PMID 24569145
- [Background] Willson JD, Petrowitz I, Butler RJ, Kernozek TW. Male and female gluteal muscle activity and lower extremity kinematics during running. Clin Biomech (Bristol). 2012 Dec;27(10):1052-7. doi: 10.1016/j.clinbiomech.2012.08.008. Epub 2012 Sep 1. PMID 22948078
- [Background] Willson JD, Davis IS. Lower extremity strength and mechanics during jumping in women with patellofemoral pain. J Sport Rehabil. 2009 Feb;18(1):76-90. doi: 10.1123/jsr.18.1.76. PMID 19321908
- [Background] Nakagawa TH, Maciel CD, Serrao FV. Trunk biomechanics and its association with hip and knee kinematics in patients with and without patellofemoral pain. Man Ther. 2015 Feb;20(1):189-93. doi: 10.1016/j.math.2014.08.013. Epub 2014 Sep 9. PMID 25261089
- [Background] Nakagawa TH, Serrao FV, Maciel CD, Powers CM. Hip and knee kinematics are associated with pain and self-reported functional status in males and females with patellofemoral pain. Int J Sports Med. 2013 Nov;34(11):997-1002. doi: 10.1055/s-0033-1334966. Epub 2013 Jun 14. PMID 23771827
- [Background] Nakagawa TH, Moriya ET, Maciel CD, Serrao FV. Trunk, pelvis, hip, and knee kinematics, hip strength, and gluteal muscle activation during a single-leg squat in males and females with and without patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2012 Jun;42(6):491-501. doi: 10.2519/jospt.2012.3987. Epub 2012 Mar 8. PMID 22402604
- [Background] Nakagawa TH, Muniz TB, Baldon RM, Maciel CD, Amorim CF, Serrao FV. Electromyographic preactivation pattern of the gluteus medius during weight-bearing functional tasks in women with and without anterior knee pain. Rev Bras Fisioter. 2011 Jan-Feb;15(1):59-65. doi: 10.1590/s1413-35552011005000003. Epub 2011 Mar 4. PMID 21390470
- [Background] Teng HL, Powers CM. Sagittal plane trunk posture influences patellofemoral joint stress during running. J Orthop Sports Phys Ther. 2014 Oct;44(10):785-92. doi: 10.2519/jospt.2014.5249. Epub 2014 Aug 25. PMID 25155651
- [Derived] Glaviano NR, Marshall AN, Mangum LC, Hart JM, Hertel J, Russell S, Saliba SA. Impairment-Based Rehabilitation With Patterned Electrical Neuromuscular Stimulation and Lower Extremity Function in Individuals With Patellofemoral Pain: A Preliminary Study. J Athl Train. 2019 Mar;54(3):255-269. doi: 10.4085/1062-6050-490-17. Epub 2019 Feb 5. PMID 30721093